CLINICAL TRIAL: NCT07068646
Title: Computed Tomogram Myocardial Thickness Map-Guided Pulmonary Vein Isolation vs. Empirical Pulmonary Vein Isolation in Pulse-Field Ablation for Paroxysmal Atrial Fibrillation (UTMOST AF III)
Brief Title: Thickness Map-Guided vs. Empirical PV Isolation Using Pulsed Field Ablation for Paroxysmal AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-0458
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT myocardial thickness map guided PV isolation group (Experimental)
  Interventions: Procedure: CT myocardial thickness map guided PV isolation group
- Empirical PV isolation group (Active Comparator)
  Interventions: Procedure: Empirical PV isolation group

INTERVENTIONS:
Procedure: CT myocardial thickness map guided PV isolation group — Pulmonary vein isolation will be performed using the PulseSelect™ pulsed field ablation system. A pre-procedural cardiac CT scan will be used to generate an atrial myocardial thickness map. In this group, atrial segments with wall thickness >2.5 mm identified on the CT map will receive additional PFA applications (up to 8 per PV) to ensure transmural lesion formation. All other segments will receive the standard minimum of 8 applications per vein. The ablation catheter will remain stationary to allow lesion stacking when needed.
  Arms: CT myocardial thickness map guided PV isolation group
Procedure: Empirical PV isolation group — Pulmonary vein isolation will be performed using the PulseSelect™ pulsed field ablation system according to a standardized empirical protocol. Each pulmonary vein will receive a minimum of 8 PFA applications without adjustment based on anatomical or CT-based parameters. Additional applications may be delivered at the operator's discretion based on procedural findings, but no wall thickness mapping will be used.
  Arms: Empirical PV isolation group

SUMMARY:
This is a prospective, multicenter, randomized controlled trial comparing CT-guided versus empirical pulsed field ablation (PFA) for pulmonary vein isolation in patients with paroxysmal atrial fibrillation. The study investigates whether atrial wall thickness-based energy titration improves arrhythmia outcomes compared to standard empirical ablation using the PulseSelect™ system.

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) using pulsed field ablation (PFA) is an effective and increasingly adopted strategy for the treatment of paroxysmal atrial fibrillation (AF). However, current empirical lesion protocols do not account for patient-specific anatomical variability, particularly atrial wall thickness, which may influence lesion durability. This randomized controlled trial aims to evaluate whether a CT-guided ablation strategy-using pre-procedural atrial wall thickness maps to titrate lesion application-can improve rhythm outcomes compared to standard empirical PFA. A total of 298 patients will be enrolled and randomized to either the CT-guided or empirical group, with follow-up over 12 months to assess freedom from atrial arrhythmia recurrence and procedure-related safety outcomes.

ELIGIBILITY:
* Patient with paroxysmal atrial fibrillation who is scheduled for ablation procedure and ≥19 and ≤80 years of age
* Left atrium size < 50mm
* paroxysmal atrial fibrillation that is recurrence during antiarrhythmic drug treatment or is not able to use an antiarrhythmic drug.
* Patient who is indicated for anticoagulation therapy (for prevention of cerebral infarction)

Exclusion Criteria:

* Patients with persistent or permanent atrial fibrillation
* Atrial fibrillation associated with severe cardiac malformation or a structural heart disease that is hemodynamically affected
* Patients with severe renal impairment or CT imaging difficulty using contrast media
* Patients with a past history of radiofrequency ablation for atrial fibrillation or other cardiac surgery
* Patients with active internal bleeding
* Patients with contraindications for anticoagulation therapy(for prevention of cerebral infarction) and antiarrhythmic drugs
* Patients with valvular atrial fibrillation (mitral stenosis >grade 2, mechanical valve, mitral valvuloplasty)
* Patients with a severe comorbid disease
* Expected survival < 1 year
* Drug addicts or alcoholics
* Patients who cannot read the consent form (illiterates, foreigners, etc.)
* Other patients who are judged by the principal or sub-investigator to be ineligible for participation in this clinical study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmia recurrence | Within 1 year after 3 months of procedure
  Any documented episode of AF, atrial flutter, or atrial tachycardia lasting ≥30 seconds after a 3-month blanking period.

SECONDARY OUTCOMES:
Procedure-related cardiac complication rate | 30 days after procedure
  Open cardiac surgery, cerebral infarction, pericardial effusion or cardiac tamponade, hematoma in the inguinal puncture site and vascular complications

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided